CLINICAL TRIAL: NCT00883844
Title: Lowering Viral Load With Nucleos(t)Ide Analogues Prior to Peginterferon Alfa-2b Treatment to Increase Sustained Response in HBeAg-positive Chronic Hepatitis B - a Pilot Study
Brief Title: PEG-IFN in HBV Patients With Incomplete Response to NA
Acronym: PADD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBV09-03
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; sustained response; peginterferon; nucleos(t)ide analogues
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Continuation of any Nucleos(t)ide analogue treatment and add-on of peginterferon for 24 weeks
  Interventions: Drug: Nucleos(t)ide analogue treatment with a peginterferon add-on strategy
- 2 (Active Comparator): Continuation of Nucleos(t)ide analogue mono-therapy
  Interventions: Drug: Nucleos(t)ide analogue treatment

INTERVENTIONS:
Drug: Nucleos(t)ide analogue treatment with a peginterferon add-on strategy — peginterferon 1.5 microgram/kg once a week Treatment with one of the approved nucleos(t)ide analogues
  Arms: 1
Drug: Nucleos(t)ide analogue treatment — Treatment with one of the approved nucleos(t)ide analogues
  Arms: 2

SUMMARY:
Treatment with a nucleoside analogue and subsequent viral decline has shown to partially restore immune hyporesponsiveness in chronic hepatitis B patients. Recent pilot studies investigating whether the effect of lowering viral load with nucleoside analogue therapy prior to the initiation of peginterferon results in higher sustained off-treatment responses showed contradictory findings.

The aim of this study is to investigate sustained off-treatment response to peginterferon alfa-2b in chronic HBeAg-positive hepatitis B patients who are pretreated with nucleos(t)ide analogues, thereby lowering viral load

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (HBsAg positive > 6 months)
* HBeAg positive, anti-HBe negative within one month prior to initiation of peginterferon alfa-2b
* HBV DNA < 2000 IU/ml during nucleos(t)ide analogue treatment within one month prior to initiation of peginterferon alfa-2b
* Compensated liver disease
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Treatment with any investigational drug within 30 days of entry to this protocol
* Severe hepatitis activity as documented by ALT>10 x ULN
* History of decompensated cirrhosis (defined as jaundice in the presence of cirrhosis, ascites, bleeding gastric or esophageal varices or encephalopathy)
* Pre-existent neutropenia (neutrophils <1,800/mm3) or thrombocytopenia (platelets <90,000/mm3)
* Co-infection with hepatitis C virus, hepatitis D virus or human immunodeficiency virus (HIV)
* Other acquired or inherited causes of liver disease: alcoholic liver disease, obesity induced liver disease, drug related liver disease, auto-immune hepatitis, hemochromatosis, Wilson's disease or alpha-1 antitrypsin deficiency
* Alpha fetoprotein > 50 ng/ml
* Hyper- or hypothyroidism (subjects requiring medication to maintain TSH levels in the normal range are eligible if all other inclusion/exclusion criteria are met)
* Immune suppressive treatment within the previous 6 months
* Contra-indications for alfa-interferon therapy like suspected hypersensitivity to interferon or Peginterferon or any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study.
* Pregnancy, breast-feeding
* Other significant medical illness that might interfere with this study: significant pulmonary dysfunction in the previous 6 months, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g. HIV positivity, auto-immune diseases, organ transplants other than cornea and hair transplant)
* Any medical condition requiring, or likely to require chronic systemic administration of steroids, during the course of the study
* Substance abuse, such as alcohol (>80 g/day), I.V. drugs and inhaled drugs in the past 2 years.
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sustained response defined as HBeAg loss and HBV DNA level < 200 IU/mL | at week 72

CONTACTS AND LOCATIONS:
Overall Officials: Harry LA Janssen, MD PhD, Principal Investigator — Erasmus MC, University Medical Center Rotterdam
Locations (2):
- Netherlands (2):
  - AMC, Amsterdam
  - Erasmus MC, University Medical Center Rotterdam, Rotterdam